CLINICAL TRIAL: NCT06142734
Title: Laparoscopic Versus Mini-incision Open Dismembered Pyeloplasty for Treatment of Ureteropelvic Junction Obstruction in Children: a Comparative Randomized Trial.
Brief Title: Laparoscopic Versus Open Pyeloplasty for Treatment of UPJO in Children.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahmed Mahmoud Abdelraouf (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mahmoud Abdelraouf, Assistant lecturer of Urology, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pyeloplasty in children
Record Dates: First submitted 2023-09-17; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Pyeloplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mini-incision open dismembered pyeloplasty (Other): Open surgery
  Interventions: Procedure: pyeloplasty
- Laparoscopic dismembered pyeloplasty (Other): Minimally invasive surgery
  Interventions: Procedure: pyeloplasty

INTERVENTIONS:
Procedure: pyeloplasty — * For laparoscopic pyeloplasty:
  * Anaesthesia: general
  * Position: a 45-degree lateral decubitus position with the concerned side up. Patient is secured to the operating table. Pneumoperitoneum is adopted through a camera port lateral to the umbilicus
  * extra operating ports are created at subcostal and at spinoumbilial line.
  * the UPJ is transperitoneally accessed by incising the white line of Toldt and the ipsilateral colon is reflected and the proximal ureter and the pelvis are identified an mobilized
  * then Anderson- Hynes pyeloplasty is carried out with insertion of nephroureterostomy or pyeloureterostomy tube.

SUMMARY:
Uretropelvic junction ( UPJ ) obstruction is a common congenital disorder , but not all cases require surgical intervention. Uretropelvic junction ( UPJ ) obstruction is a common congenital disorder , but not all cases require surgical intervention. On the other hand, in children many authors reported mini incision open pyeloplasty with very small subcostal muscle splitting incision, with negligible postoperative pain and very short hospital stay

DETAILED DESCRIPTION:
Uretropelvic junction ( UPJ ) obstruction is a common congenital disorder , but not all cases require surgical intervention. Indications for surgical intervention include impaired split renal function (< 40%), a decrease of split renal function of > 10% in subsequent studies, poor drainage function after the administration of furosemide, increased anteroposterior diameter on US, and grade III and IV dilatation as defined by the Society for Fetal Urology. The open dismembered pyeloplasty was the historical gold standard repair of uretropelvic junction obstruction. Schuessler et al. introduced the first laparoscopic pyeloplasty (LP) 1993 followed by Peters et al, who performed the first pediatric laparoscopic pyeloplasty. Since then, minimally invasive pyeloplasty (MIP) -laparoscopic and robotic assisted- had an increasing interest among urologists and became widely adopted by many centers as a standard surgical intervention in UPJ obstruction; thanks to the decreased postoperative pain, short hospital stay, reduced postoperative recovery time, and comparable success rates. The high cost and long learning curve hindered generalization of MIP in all centers. On the other hand, in children many authors reported mini incision open pyeloplasty with very small subcostal muscle splitting incision, with negligible postoperative pain and very short hospital stay . Tanaka et al. have reported that the benefits of laparoscopic pyeloplasty were evident only in older children . Till now 85% of infants are still treated with open pyeloplasty . According to the EAU guidelines 2023 "There does not seem to be any clear benefit of minimally invasive procedures in a very young child but current data are insufficient to defer a cut-off age " .

Most of the studies that compared open to LP didn't limit cases to mini-incision open pyeloplasty.

To our knowledge there is no prospective randomized study comparing laparoscopic to open pyeloplasty with mini-incision in children to date.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1-18 years , males and females with UPJ obstruction in orthotopic kidney indicated for dismembered pyeloplasty and not else

Exclusion Criteria:

* Recurrent UPJ obstruction.
* Cases that require technique other than dismembered pyeloplasty
* Patients that have contradiction to laparoscopy.
* comorbidities that prevent surgery e.g: uncorrected coagulopathy and vertebro-spinal deformity
* patient refusing participation in the study.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Operative time | baseline
  From incision to last stitch